CLINICAL TRIAL: NCT06427226
Title: Clinical Study to Evaluate the Possible Safety and Efficacy of Dapagliflozin in the Prophylaxis of Doxorubicin-Induced Cardiotoxicity in Breast Cancer Patients
Brief Title: Evaluation of the Possible Safety and Efficacy of Dapagliflozin in the Prophylaxis of Doxorubicin-Induced Cardiotoxicity
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sandy Ehab Nabil Rezkallah, Clinical Pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dapagliflozin in breast cancer
Record Dates: First submitted 2024-05-18; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Doxorubicin Induced Cardiomyopathy; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — dapagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): 23 breast cancer patients which will receive four cycles of AC regimen (Doxorubicin and Cyclophosamide; each cycle is given every 21 days) only.
- Dapagliflozin group (Active Comparator): 23 breast cancer patients which will receive four cycles of AC regimen (Doxorubicin and Cyclophosamide; each cycle is given every 21 days) plus Dapagliflozin 10 mg once daily.
  Interventions: Drug: Dapagliflozin 10mg Tab

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin 10 mg tab once daily given during the duration of AC cycles.
  Arms: Dapagliflozin group

SUMMARY:
This is a randomized controlled clinical trial that aims to evaluate the safety and efficacy of Dapagliflozin as a cardioprotective in doxorubicin-induced cardiotoxicity in breast cancer patients.

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer in women and the first cause of cancer death among them. In Egypt, it represents 33%of female cancer cases and more than 22,000 new cases are diagnosed each year. This is expected to rise exponentially over the next years given the enlarging population and changes in the population pyramid.

The Early Breast Cancer "Trialists" Collaborative Group (EBCTCG) reported that the inclusion of anthracyclines as doxorubicin in the management of breast cancer improved absolute survival by approximately 3% at 5 years and 4% at 10 years. Therefore, anthracyclines remain the cornerstone of treatment for breast cancer patients.

Despite its effectiveness, doxorubicin is associated with cumulative, dose-dependent, and potential cardiotoxicity.

Although the main mechanism of doxorubicin-induced cardiotoxicity has not been fully known, there are several mechanisms proposed for cardiac injury including oxidative stress, free radical generation, and apoptosis are most widely reported. Other mechanisms are also involved such as impaired mitochondrial function, perturbation in iron regulatory protein, disruption of Ca2+ homeostasis, autophagy, and the release of nitric oxide and inflammatory mediators.

Dapagliflozin (DAPA), a sodium-glucose cotransporter 2 (SGLT2) inhibitor, is a class of glucose-lowering agents and is used to treat patients with type 2 diabetes. Besides reducing glucose reabsorption, DAPA has shown protective effects on cardiovascular diseases. The cardioprotective effects of DAPA have been demonstrated in patients with diabetic cardiomyopathy, heart failure (HF) with preserved ejection fraction (EF), and HF with reduced EF. SGLT2 inhibitors exert their cardioprotective effect by increasing energy metabolism, mitochondrial biogenesis, autophagy, and ketone bodies while decreasing endoplasmic reticulum (ER) stress, ferroptosis, oxidative stress, and inflammation.

In a recent animal study, DAPA protected against doxorubicin-induced cardiotoxicity by reducing ER stress, as evidenced by the decreased expression of the ER-related proteins including glucose-regulated protein 78, protein kinase R-like endoplasmic reticulum kinase and transcription factor 4.

Doxorubicin administration have been shown to increase HF incidence, HF admissions, and the development of cardiomyopathy which is defined by a decline in left ventricle ejection fraction and these outcomes were attenuated by SGLT2 inhibitors.

It is known that doxorubicin increases the circulating level of N-terminal pro-B-type natriuretic peptide (NT-pro-BNP) and cardiac Troponin T (cTnT) which DAPA significantly reduced in a recent animal study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Chemo-naïve patients with biopsy confirmed diagnosis of breast cancer and with stage I-III breast cancer according to the American Joint Committee on Cancer (TNM staging system of breast cancer).
* Patients intended to receive at least 4 cycles of doxorubicin or more.
* Patients with performance status <2 according to Eastern Cooperative Oncology Group (ECOG) score.
* Echocardiographic LVEF ≥55%.
* Adequate baseline hematologic values (absolute neutrophilic count ≥ 1.5 ×109/L, platelet count ≥ 90 × 109/L and hemoglobin level ≥ 10 g/dl).
* Patients with adequate liver function and adequate renal function.
* Signed informed consent to participate in the study.

Exclusion Criteria:

* Age <18 years old and >65 years old.
* Patients with prior exposure to anthracyclines within the last 6 months.
* Patients with evidence of metastasis at initial assessment.
* Treatment with any SGLT-2 inhibitors for 6 months prior to the screening.
* Patients taking any other cardioprotective medications.
* Pregnancy and breast feeding.
* Alcohol abuse.
* History of heart failure or LVEF <50%.
* Presence of any cardiac-related conditions such as angina pectoris, valvular disease, uncontrolled systemic hypertension, coronary heart disease, and cardiac surgery within the last 3 months.
* Patients with type 1 diabetes mellitus or diabetic ketoacidosis, history of stroke, and patients with severe renal impairment with GFR <25ml/min/1.73m2 . - Patients taking gatifloxacin as it causes major drug interaction with dapagliflozin.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer patients
Enrollment: 46 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of changes in ejection fraction using echocardiography | Baseline and after the last AC cycle of chemotherapy (3months).
  Initial evaluation of cardiac function by Echocardiography at baseline and after the end of chemotherapy. The primary outcome is to avoid reduction in patients' ejection fraction during doxorubicin administration.

SECONDARY OUTCOMES:
Change in Cardiac Troponin T level | Baseline and after the last AC cycle of chemotherapy (3months).
  Monitoring the serum biomarker Cardiac Troponin T at baseline and after the end of chemotherapy.
Change in N-terminal pro-B-type natriuretic peptide level | Baseline and after the last AC cycle of chemotherapy (3months).
  Monitoring the serum biomarker NT-pro-BNP at baseline and after the end of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Sandy E Rezkallah, bachelor, Principal Investigator — Tanta University
Locations (1):
- Medical Research Institute, Alexandria, Bab Sharqi, Egypt

REFERENCES:
- [Background] Belen E, Canbolat IP, Yigitturk G, Cetinarslan O, Akdeniz CS, Karaca M, Sonmez M, Erbas O. Cardio-protective effect of dapagliflozin against doxorubicin induced cardiomyopathy in rats. Eur Rev Med Pharmacol Sci. 2022 Jun;26(12):4403-4408. doi: 10.26355/eurrev_202206_29079. PMID 35776041
- [Background] Avula V, Sharma G, Kosiborod MN, Vaduganathan M, Neilan TG, Lopez T, Dent S, Baldassarre L, Scherrer-Crosbie M, Barac A, Liu J, Deswal A, Khadke S, Yang EH, Ky B, Lenihan D, Nohria A, Dani SS, Ganatra S. SGLT2 Inhibitor Use and Risk of Clinical Events in Patients With Cancer Therapy-Related Cardiac Dysfunction. JACC Heart Fail. 2024 Jan;12(1):67-78. doi: 10.1016/j.jchf.2023.08.026. Epub 2023 Oct 25. PMID 37897456
- [Background] Chang WT, Lin YW, Ho CH, Chen ZC, Liu PY, Shih JY. Dapagliflozin suppresses ER stress and protects doxorubicin-induced cardiotoxicity in breast cancer patients. Arch Toxicol. 2021 Feb;95(2):659-671. doi: 10.1007/s00204-020-02951-8. Epub 2020 Nov 19. PMID 33211168